CLINICAL TRIAL: NCT00124696
Title: Cocaethylene Substitution Therapy and Tolerance Induction in Treating Cocaine Dependence
Brief Title: Cocaethylene as a Treatment for Cocaine Dependence - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-13586-1; R01-13586-1; DPMC
Record Dates: First submitted 2005-07-22; First posted 2005-07-28 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2005-08

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — cocaethylene

INTERVENTIONS:
Drug: Cocaethylene

SUMMARY:
Cocaine has been cited as the primary drug threat in the United States. The purpose of this study is to determine if cocaethylene, used as a prototype drug, is a safe and effective treatment for cocaine dependence.

DETAILED DESCRIPTION:
Currently, there are no medications available to specifically treat cocaine addiction. Cocaethylene is an active metabolite of cocaine and has a similar chemical structure to cocaine. The purpose of this study is to determine whether substitution therapy with cocaethylene is a safe and effective treatment for cocaine dependence.

This double-blind, placebo-controlled trial will occur in 3 parts. In Part 1, the individual pharmacokinetics of an intravenous dose of cocaethylene will be determined in order to estimate individualized cocaethylene infusion rates and pharmacokinetic parameters. This will provide important information on how cocaethylene is processed by the body. In Part 2, an infusion of cocaethylene, producing a venous plasma concentration of 200 ng/ml, will be administered over an 8-hour period. Clinical monitoring and blood sampling will occur in order to determine the safety profile of cocaethylene. During Part 3, the ability of cocaethylene to modify the acute effects of intravenous cocaine will be determined. Cocaethylene will be administered in plasma concentrations of 0 ng/ml, 50 ng/ml, or 200 ng/ml over an 8-hour period. Participants will be randomly assigned to receive a challenge intravenous dose of cocaine (0.5 mg/kg or 1 mg/kg) or placebo at the 4-hour mark of cocaethylene infusion. Following the initial 8-hour period, cocaethylene infusion will be continued for an additional 5 hours. Behavioral and physiological measures will be collected throughout the study sessions at predetermined times to evaluate whether tolerance to cocaethylene develops. These measures will also help to determine whether cocaethylene modifies or produces tolerance to the effects of an acute dose of cocaine.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for cocaine dependence
* Cocaine use of at least 0.5 grams each week during the three months prior to enrollment, confirmed by a positive urine test for cocaine metabolite
* Females are eligible if currently using adequate contraception, not planning to become pregnant, or surgically sterilized
* Females of child-bearing potential must have a negative pregnancy test prior to study entry
* Currently not physiologically dependent on alcohol, but may meet DSM-IV criteria for alcohol abuse or dependence

Exclusion Criteria:

* Meets DSM-IV criteria for dependence on any drugs (other than nicotine or alcohol) within the year prior to enrollment
* Currently abuses other substances such as opiates, sedative-hypnotics, or amphetamines (excluding marijuana or nicotine) more than twice a week
* History of a serious medical illness or indication of a serious medical illness such as seizures, hypertension, heart disease, an abnormal ECG, anemia, diabetes, or abnormal blood flow sounds
* Meets DSM-IV criteria for a current major mental disorder, including major depression, bipolar disorder, schizophrenia, schizophreniform disorder, schizoaffective disorder, mental retardation, or organic mental syndrome
* Currently being treated with psychotropic medication
* At risk for suicide, as determined by a psychiatrist
* Greater than two times the normal level for liver or kidney function tests
* Currently seeking treatment for drug abuse
* Participants with liver function tests equal to or greater than three times the normal level will be discontinued from the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8
Dates: Start 2002-12; Study Completion 2005-03

PRIMARY OUTCOMES:
Clinical physiological response to cocaine challenge - especially adverse effects measures

CONTACTS AND LOCATIONS:
Overall Officials: Elinore Mccance-Katz, M.D., Ph.D., Principal Investigator — Yale Psychiatric Institute
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States